CLINICAL TRIAL: NCT03956459
Title: Evaluation of PET-CT Scanner Performances to Detect Infra-centimetric Lesions in Patients With Cancer
Acronym: IQversusMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19 GENE 03
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cancer
Keywords: FDG-PET
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a cancer (Other)
  Interventions: Other: Patients with a cancer for which a FDG-PET scanner must be performed

INTERVENTIONS:
Other: Patients with a cancer for which a FDG-PET scanner must be performed — For each patient, 2 consecutive PET-CT scanners will be performed using 2 different systems of PET-CT scanners:
  * "Discovery MI"
  * "Discovery IQ"
  Only one contrast agent injection (FDG) will be given for both scanners.

SUMMARY:
Prospective, monocentric study aiming to evaluate the PET-CT (Positron Emission Tomography - Computed Tomography) scanner performances to detect infra-centimetric lesions in two groups of patients with cancer and of different BMI (Body Mass Index) classes (BMI ≤ 25 and BMI > 25).

For each patient, two consecutive PET-CT scanner will be performed using the "Discovery MI" and "Discovery IQ" PET-CT scanner systems.

Virtual lesions will then be created on images obtained. Images will be interpreted by two independent observers.

The study participation of each patient will be a maximum of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. A patient with a cancer for which a FDG-PET (fluorodeoxyglucose-positron emission tomography) must be performed according to the standard practices
3. OMS ≤ 1, Karnofsky Index > 70.
4. Negative pregnancy test at inclusion.
5. Patient able to maintain a lying position in a strict supine position twice.
6. Patient affiliated to a Social Health Insurance in France.
7. Patient who has signed informed consent prior inclusion in the study and before any specific procedures for the study.

Exclusion Criteria:

1. Patient with unbalanced diabetic
2. Patient with a formal contraindication usual for certain imaging procedures (severe claustrophobia, wearing a heart valve, pacemaker, etc.)
3. Pregnant or breastfeeding woman
4. Any psychological, family, geographical or sociological condition that does not allow medical follow-up and/or procedures provided for in the study protocol to be respected
5. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Relative rate of virtual lesions detected by each system ("Discovery MI" and "Discovery IQ") | 24 hours for each patient

SECONDARY OUTCOMES:
Rate of Inter-observer concordance in radiological images interpretation | 24 hours for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse, France